CLINICAL TRIAL: NCT03230188
Title: Patterns of Neurocircuitry Activation In Severe Asthma
Acronym: PANISA
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2017-0208; 5R01HL123284-02 (NIH)
Record Dates: First submitted 2017-06-28; First posted 2017-07-26 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Lung Diseases
Keywords: asthma; neurocircuitry; severe asthma; mild to moderate asthma; neurocircuitry patterns
MeSH Terms: conditions — Lung Diseases; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe Asthmatics: Individuals with severe asthma that are already enrolled in the University of Wisconsin Severe Asthma Research Program III study will fill out asthma and psychological questionnaires (non-diagnostic), will undergo Cognitive Function Testing (non-diagnostic), and will undergo a simulated and actual functional Magnetic Resonance Imaging (research grade) scan.
  Interventions: Other: functional Magnetic Resonance Imaging (research grade); Other: Cognitive Function Testing (non-diagnostic); Other: Asthma and Psychological Questionnaires (non-diagnostic)

INTERVENTIONS:
Other: functional Magnetic Resonance Imaging (research grade) — Subjects will undergo a simulated and actual functional Magnetic Resonance Imaging scan.
Other: Cognitive Function Testing (non-diagnostic) — Subjects will take non-diagnostic cognitive function tests
Other: Asthma and Psychological Questionnaires (non-diagnostic) — Subjects will fill out asthma and psychological questionnaires (non-diagnostic)

SUMMARY:
The overall purpose of the study is to compare the patterns of neurocircuitry activation in severe asthmatics vs. mild to moderate and healthy controls. The Investigators hypothesize that neurocircuitry activation increases with asthma severity, producing different neurocircuitry patterns for severe asthmatics than those of mild to moderate asthmatics or non-asthmatics.

DETAILED DESCRIPTION:
To begin to further address possible relationships of asthma and brain function, the investigators propose the following hypothesis, "patients with defined characteristics of severe asthma will have distinct patterns of persistent neurocircuitry activation. The investigators further propose that the detection of ongoing neurocircuitry activation occurs because of persistent and active airway inflammation in severe asthma. Finally, the investigators propose that the intensity of specific neurocircuitry activation will relate to the severity of underlying asthma.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in Severe Asthma Research Program III (2012-0571) study
* Has severe asthma
* Is a male or female with no health concerns that might affect the outcome of the study
* Provided a negative urine pregnancy test prior to visit (Females only)
* Capable and willing to grant written informed consent and cooperate with study procedures and requirements (investigator discretion)
* Is able to tolerate a simulated functional Magnetic Resonance Imaging brain scanning session
* Is able to give valid informed consent to participate by signing and dating a written consent form

Exclusion Criteria:

* Uses psychotropic medication that might affect function of neurocircuitry implicated in our hypotheses (at the discretion of a study physician or Co-Investigator)
* Has one or more contraindications for functional Magnetic Resonance Imaging
* Has needle phobia or claustrophobia
* Unable to distinguish specific colors used in Stroop task
* History of a diagnosed Bipolar Disorder, Schizophrenia, or Schizoaffective Disorder
* Is a pregnant or lactating female
* Has had an upper or lower respiratory infection within 1 month of the visit
* Has unstable asthma as indicated by self-report of increased symptoms or increased beta-agonist use over the 2 weeks preceding the visit
* Is a current smoker (defined as smoked within the last year) or a former smoker with a history of >5 pack years
* Any condition which, in the opinion of the investigator, might interfere with participation in the study
* Inability or unwillingness to perform required study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults ages 18 and older who are currently rolled in the Severe Asthma Research Program III study at the University of Wisconsin-Madison (all subjects have severe asthma)
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-17 (Actual); Study Completion 2018-06-17 (Actual)

PRIMARY OUTCOMES:
Measures of Neural Activity | Visit 1 (1 day)
  % signal change in brain insula detected by functional Magnetic Resonance Imaging

SECONDARY OUTCOMES:
Airway Cellular and Molecular Inflammatory Response- White Blood Cells | Visit 1 (1 day)
  Cell differential counts- Total White Blood Cell count (sum of absolute counts for: Eosinophils, Monocytes, Neutrophils, Basophils, Lymphocytes)
Airway Cellular and Molecular Inflammatory Response- Eosinophils | Visit 1 (1 day)
  Cell differential counts- Eosinophils
Airway Cellular and Molecular Inflammatory Response- Lymphocytes | Visit 1 (1 day)
  Cell differential counts- Lymphocytes (absolute lymphocyte count, percent lymphocytes)
Airway Cellular and Molecular Inflammatory Response- Monocytes/Macrophages | Visit 1 (1 day)
  Cell differential counts- Monocytes/Macrophages (absolute monocyte count, percent monocytes)
Airway Cellular and Molecular Inflammatory Response- Neutrophils | Visit 1 (1 day)
  Cell differential counts- Neutrophils (absolute neutrophil count, percent neutrophils)

CONTACTS AND LOCATIONS:
Overall Officials: William W Busse, MD, Principal Investigator — The University of Wisconsin School of Medicine and Public Health
Locations (1):
- UW Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT03230188/Prot_SAP_003.pdf